CLINICAL TRIAL: NCT01042145
Title: Community Care for Croup (RCT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Washington University Pediatric and Adolescent Ambulatory Research Consortium (Network)
Responsible Party: Principal Investigator, Jane Garbutt, MD, Associate Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09-0542; NIH/NCRR UL1RR024992
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Croup
Keywords: Primary Care; Treatment; Croup; Corticosteroids; Prednisone; Dexamethasone; Randomized trial
MeSH Terms: conditions — Croup | interventions — Prednisone; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisone (Active Comparator): Prednisone, 2mg/kg for 3 days
  Interventions: Drug: Prednisone
- Dexamethasone (Active Comparator): Dexamethasone, 0.6mg/kg for one day, then placebo for 2 days
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Prednisone — 2 mgs/kg for 3 days
  Arms: Prednisone
Drug: Dexamethasone — 0.6 mgs for one day, then placebo for 2 days
  Arms: Dexamethasone

SUMMARY:
This randomized clinical trial was to compare the effectiveness of prednisone 2mg/kg/day for 3 days vs. dexamethasone 0.6mg/kg for 1 day for treatment of children with mild or moderate croup. It was conducted in a practice-based research network of community pediatricians in the St. Louis area. Outcomes included additional health care for croup, duration of symptoms, nights of disturbed sleep, parental stress, missed work days, and adverse events. Our hypothesis was that community-based treatment of children with mild or moderate croup with multiple doses of prednisone is superior to a single dose of dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* children aged 1 to 8 years old (not yet reached their 9th birthday), who have croup symptoms for less than or equal to 48 hours and have a physician diagnosis of mild or moderate croup.

Exclusion Criteria:

* Severe croup or impending respiratory failure;
* another reason to indicate the need for hospitalization;
* symptoms or signs to suggest another cause of stridor;
* active varicella infection;
* diabetes;
* known immunodeficiency disease;
* chronic respiratory disease such as CF (Cystic Fibrosis);
* prescribed a controller medication or oral steroids for asthma in the past 12 months;
* a history of TB(tuberculosis) in a household member;
* treatment for seizures;
* treatment with epinephrine or oral corticosteroids for this croup episode before enrollment;
* not accompanied by their legal guardian;
* the accompanying adult will not be in the same household as the child for the next four days;
* parent/legal guardian is unavailable for telephone follow-up or does not speak English.

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2009-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane M Garbutt, MB, ChB, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Result] Garbutt JM, Conlon B, Sterkel R, Baty J, Schechtman KB, Mandrell K, Leege E, Gentry S, Stunk RC. The comparative effectiveness of prednisolone and dexamethasone for children with croup: a community-based randomized trial. Clin Pediatr (Phila). 2013 Nov;52(11):1014-21. doi: 10.1177/0009922813504823. Epub 2013 Oct 3. PMID 24092872

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children were recruited from 10 primary care pediatric practices over two winters: between October 26, 2009 and April 16, 2010; and between September 6, 2010 and April 29, 2011.
Pre-assignment Details: 103 children were assessed for eligibility. 16 were excluded prior to randomization. reasons were: did not meet inclusion criteria (10), declined to participte (6).
Period: Overall Study
Arm/Group | Prednisone | Dexamethasone
Started | 41 | 46
Completed | 40 | 45
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prednisone | Dexamethasone | Total
Number analyzed (Participants) | 41 | 46 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 41 | 46 | 87
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.67 (1.43) | 3.11 (1.58) | 2.9 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 18 | 31
  Male | 28 | 28 | 56
Region of Enrollment [Number; unit: participants]
  United States | 41 | 46 | 87

OUTCOME MEASURES:

1. Primary Outcome: Additional Health Care
Description: The primary outcome was the % of participants who had additional health care for croup within 11 days of randomization assessed by self-report. This dichotomous variable was positive if any of the following occurred: office visit, ED visit or hospitalization for croup care.
Time Frame: 11 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prednisone | Dexamethasone
Number analyzed (Participants) | 40 | 45
percentage of participants | 7 [1.5 to 19.9] | 2 [0 to 11.5]
Statistical Analysis 1: Comparison: Prednisone vs Dexamethasone; Test type: Superiority or Other; p = 0.34, Fisher Exact

2. Secondary Outcome: Duration of Croup Symptoms
Time Frame: 12 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Prednisone | Dexamethasone
Number analyzed (Participants) | 40 | 45
days | 2.2 (1.3) | 2.8 (2.7)
Statistical Analysis 1: Comparison: Prednisone vs Dexamethasone; Test type: Superiority or Other; p = 0.63, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Nights With Disturbed Sleep
Time Frame: 12 days
Measure: Mean (Standard Deviation); unit: nights
Arm/Group | Prednisone | Dexamethasone
Number analyzed (Participants) | 40 | 45
nights | 1.21 (2.69) | 0.68 (1.55)

4. Secondary Outcome: Parental Stress
Description: Parental stress due to the child's illness was rated using a 4-point categorical scale (ranging from 3-very stressed to 0-not stressed). We report days until the stress rating was 0.
Time Frame: 12 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Prednisone | Dexamethasone
Number analyzed (Participants) | 40 | 45
days | 1.56 (2.69) | 1.39 (1.08)
Statistical Analysis 1: Comparison: Prednisone vs Dexamethasone; Test type: Superiority or Other; p = 0.51, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Time Missed From Work
Time Frame: 12 days
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Prednisone | Dexamethasone
Number analyzed (Participants) | 40 | 45
Hours | 3.79 (7.40) | 4.06 (5.54)
Statistical Analysis 1: Comparison: Prednisone vs Dexamethasone; Test type: Superiority or Other; p = 0.24, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Participants With Reported Side Effects
Time Frame: 12 days
Measure: Number; unit: percentage of participants
Arm/Group | Prednisone | Dexamethasone
Number analyzed (Participants) | 40 | 45
percentage of participants | 26 | 24
Statistical Analysis 1: Comparison: Prednisone vs Dexamethasone; Test type: Superiority or Other; p = 1.0, Fisher Exact

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Prednisone | Dexamethasone
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/46
Other Adverse Events (participants affected / at risk) | 0/41 | 0/46

LIMITATIONS AND CAVEATS:
Our failure to demonstrate any difference bewteen the two study groups may be due to the small sample size. We were unable to recruit the targeted sample size of 200.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes